CLINICAL TRIAL: NCT01763879
Title: Right Ventricular Function During One-lung Ventilation: The Effects of Pressure Controlled and Volume Controlled Ventilation
Brief Title: Pressure-controlled vs Volume Controlled Ventilation on RV Function During OLV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2012081; 2012081 (Other Grant/Funding Number: University of Dammam)
Record Dates: First submitted 2012-12-30; First posted 2013-01-09 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Lung Diseases
Keywords: Thoracic surgery; one lung ventilation; pressure-controlled ventilation; volume-controlled ventilation; right ventricular function
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The PCV-VCV group (Active Comparator): The dependent lung will be ventilated with pressure controlled (PCV) followed by the volume-controlled ventilation (VCV)
  Interventions: Other: The PCV-VCV group
- The VCV-PCV group (Active Comparator): The dependent lung will be ventilated with volume-controlled ventilation (VCV) followed by the pressure controlled (PCV)
  Interventions: Other: The VCV-PCV group

INTERVENTIONS:
Other: The PCV-VCV group — During the PCV period, the inspiratory pressure will be adjusted to deliver a TV of 6 mL/kg (predicted body weight) to the patient's dependent lung. During the VCV period, the patient's dependent lung will be ventilated with a TV of 6 mL/kg (PBW). Whereas FiO2, I: E ratio, PEEP, frequency, Ppk, and a FGF will be maintained as during two-lung ventilation (TLV) and the lumen of the nondependent lung will be left open to air. Dependent lung recruitment maneuvers will be repeated at 30-minute intervals by raising the inspiratory pressure up to 35 cmH2O for 10 seconds.
  Arms: The PCV-VCV group
Other: The VCV-PCV group — During the PCV period, the inspiratory pressure will be adjusted to deliver a TV of 6 mL/kg (predicted body weight) to the patient's dependent lung. During the VCV period, the patient's dependent lung will be ventilated with a TV of 6 mL/kg (PBW). Whereas FiO2, I: E ratio, PEEP, frequency, Ppk, and a FGF will be maintained as during two-lung ventilation (TLV) and the lumen of the nondependent lung will be left open to air. Dependent lung recruitment maneuvers will be repeated at 30-minute intervals by raising the inspiratory pressure up to 35 cmH2O for 10 seconds.
  Arms: The VCV-PCV group

SUMMARY:
The use of pressure controlled ventilation (TV) during one lung ventilation (OLV) for thoracic surgery is associated with comparable oxygenation with volume controlled ventilation (VCV) with added benefits of decreasing airway pressures and shunt fraction. The later may improve the right ventricular (RV) function during OLV. We postulate that the use of PCV during OLV for thoracic surgery would preserve RV function than during VCV. After local ethics committee approval and informed consent, we will randomly allocate 28 patients scheduled for elective thoracic surgery OLV to randomly crossed from PCV to VCV mode (n= 14 for each) during with VT of 6 mL/kg, I: E ratio 1: 2.5, PEEP of 5 cm H2O, recruitment maneuvers and respiratory rate will be adjusted to maintain normocapnia. Intraoperative changes in the right ventricular function (peak systolic and diastolic tricuspid annular velocity (TAV), end-diastolic volume (EDV), end-systolic volume (ESV), and RV fractional area changes (RV-FAC)), hemodynamic and oxygenation parameters, peak and plateau airway pressures, compliance will be recorded.

DETAILED DESCRIPTION:
One-lung ventilation (OLV) provides excellent operative field for thoracic procedures, but is opposed by the harmful impairment of cardiac index and right ventricular (RV) function which may influence postoperative morbidity and mortality. In our previous study, we demonstrated significant reductions in RV ejection fraction (REF) and CI values after the initiation of OLV attributable to the increased right ventricular afterload, stroke work and end-diastolic volume augmented by increased airway pressures. This may be harmful with the patients with advanced obstructive lung diseases and those with pulmonary hypertension. Thus there is no doubt that decreases in airway pressures will be associated with better RV function.

Volume controlled ventilation (VCV) is the commonly used traditional ventilation mode for OLV during thoracic procedures but its use is associated with deleterious increases in airway pressure which may impede RV function.

Pressure controlled ventilation (PCV) is an alternative mode of ventilation which is widely used in the patients with acute respiratory distress syndrome (ARDS) and acute lung injury (ALI), whereby high initial flow rates are delivered to quickly achieve and maintain the set inspiratory pressure followed by rapidly decelerating flow.These high initial flow rates lead to a more rapid alveolar inflation.

PCV has been suggested as a useful tool to improve oxygenation as well as decreases in intra-pulmonary shunt (Qs/Qt) and airway pressures compared with VCV during OLV for patients undergoing thoracic surgery. Whereas, others demonstrated comparable arterial oxygenation with the use of PCV and VCV during OLV.

However, the use of PCV offers advantages over VCV during OLV in the term of reducing mean and bronchial peak airway pressures and intrapulmonary shunt, hence limiting the risk for barotrauma and impaired RV function.

Up to the investigators knowledge, there is no available study of the effects of PCV and VCV on RV function during OLV after thoracic surgery.

The investigators hypothesize that the use of PCV during OLV will be associated with preserved RV function than during the use of VCV. They will compare the effects of the use of PCV and VCV with 5 cm H2O level of PEEP and recruitment maneuvers during OLV on the right ventricular function (peak systolic and diastolic tricuspid annular velocity (TAV), end-diastolic volume (EDV), end-systolic volume (ESV), and RV fractional area changes (RV-FAC)), hemodynamic parameters (heart rate (HR), mean arterial blood pressure, (MAP)), oxygenation parameters (arterial oxygen and carbon dioxide tension (PaO2 and PaCO2, respectively), and arterial tension to inspired fraction of oxygen (PaO2/FiO2) ratio), ventilation parameters (peak and plateau airway pressures (Ppk and Ppl, respectively) and compliance) and the ICU and hospital length-of-stays, morbidity and 30-day mortality.

Sample size calculation:

A priori power analysis of the previous published data11 showed that the investigators will need to study 13 pairs to detect a 20% difference in the mean maximal systolic TAV values (7.0 cm/s) with a SD of 1.4 cm/s, after start of OLV, a type-I error of 0.05 and a power of 90%. We will add 10% more patients for a final sample size of 28 patients to account for patients dropping out during the study.

Interventions:

In all patients, standard monitors will be applied. A thoracic epidural or paravertebral catheter will be inserted with no more use of local anesthetics during the study to avoid their effects on hypoxic pulmonary vasoconstriction.12 An arterial line (20 G) and a right internal jugular vein catheter will be inserted. Anesthetic technique will be standardized in all studied patients. Anesthesiologists who will give the anaesthetic will be not involved in the patient's assessment. General anesthesia will be induced with propofol (2-3 mg/kg), fentanyl (2-3 µg/kg), and cisatracurium (0.2 mg/kg) will be given to facilitate tracheal intubation with a left-sided double-lumen tube (DLT). The correct position of its tip will be confirmed with a fiberoptic bronchoscope. Anesthesia will be maintained with 1-1.5 minimum alveolar concentration (MAC) of sevoflurane and increments of fentanyl (0.5µg/kg) and cisatracurium (0.04 mg/kg).

The patients' lungs will be mechanically ventilated using VCV mode, fraction of inspired oxygen (FiO2) of 0.5 in air, tidal volume (VT) of 8 mL/kg (predicted body weight), inspiratory to expiratory [I: E] ratio of 1:2.5, a positive end-expiratory pressure (PEEP) of 5 cm H2O, respiratory rate (R.R) will be adjusted to achieve an PaCO2 of 35-45 mm Hg, peak inspiratory pressures (Ppk) will be limited to 35 cm H2O and a low fresh gas flow (FGF) (<2 L/min) in a semi closed circuit system.

Transesophageal echocardiography (TEE) will be inserted and the right ventricular function will be assessed with the measurements of EDV, ESV, RVEF, both maximal systolic and diastolic TAV at the tricuspid annulus at the RV free wall recorded from the apical 4-chamber views using pulsed wave Doppler tissue imaging.

All operations will be performed by the same surgeons. Intraoperative hypoxemia will be defined as decrease in arterial oxygen saturation less than 90% will be treated with increasing of FiO2 to 1.0. Addition of low level of 2 cm H2O of CPAP will be considered if the later fails to correct hypoxemia. 1 Intraoperative fluid therapy will include intravenous infusion of 2 ml/kg/hour of Lactated Ringer's solution and blood losses will be compensated with colloids and with red blood cell concentrates if the hemoglobin levels decreases below 8 to 9 g/dL. Mean arterial blood pressure will be maintained greater than 60 mm Hg using bolus doses of ephedrine 5 mg or phenylephrine 100 ug. Urine output will be maintained to be greater than 0.5 ml/kg/hour.

At the end of surgery, the nondependent will be re-expanded and TLV will be resumed as before surgery, sevoflurane will be discontinued, the residual neuromuscular block will be antagonized, and the patient will be extubated. Postoperative analgesia will be accomplished with the use of continuous epidural/paravertebral infusion of bupivacaine 0.125% and fentanyl 2 µg/mL.

Statistical Analysis:

Data will be tested for normality using the Kolmogorov-Smirnov test. Fisher exact test will be used for categorical data. Repeated two-way ANOVA and paired t-test will be used to study the changes in the primary and secondary endpoints during each intervention. The Wilcoxon 2 rank sum test will be used for the non-parametric values. We will avoid the carryover effect (persistence of the effect of the first intervention on the operative conditions into the second period) through the comparison of the effects of period (time effect) and the order of treatment using independent t-tests. Data will be expressed as mean ± SD, number (%), or median [range]. A value of P < 0.05 will be considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical class from II to III

Exclusion Criteria:

* decompensated cardiac (New York Heart Association >II)
* pulmonary (vital capacity or FEV1% < 50% of the predicted values)
* asthma
* hepatic diseases.
* renal diseases
* arrhythmias
* pulmonary hypertension (mean pulmonary artery pressure >30 mm Hg)
* body mass index >35 kg/m2
* previous history of pneumonectomy, bilobectomy, or lobectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Right ventricular function | Change from baseline at 30 min after the initiation of the intervention
  Peak systolic and diastolic tricuspid annular velocity (TAV)

SECONDARY OUTCOMES:
Blood pressure | Change from baseline at 30 min after the initiation of the intervention
  Blood pressure
Pa/FiO2 ratio | Change from baseline at 30 min after the initiation of the intervention
  the ratio between arterial oxygen tension (PaO2)and inspired fraction of oxygen (FiO2)
Airway pressures | Change from baseline at 30 min after the initiation of the intervention
  Peak and plateau airway pressures
Right ventricular volumes | Change from baseline at 30 min after the initiation of the intervention
  right ventricular end diastolic and systolic volumes

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, MD, Study Director — Assistant Professor; Roshdi Al Metwally, MD, Principal Investigator — Associate Professor; Hatem Qutub, MD, Study Chair — Associate Professor; Yasser F El Ghoneimy, MD, Study Chair — Associate Professor; Mohamed A Regal, MD, Study Chair — Associate Professor; Haytham Zien, MD, Study Chair — Assistant Professor
Locations (1):
- Anesthesiology Department, Khobar, Eastern Province, Saudi Arabia